CLINICAL TRIAL: NCT03720925
Title: Evaluation of a Dental Trauma Care Program on the Oral Health-related Quality of Life in Children and Their Families
Brief Title: Traumatic Dental Injuries Treatment and Oral Health Related to Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Livia Azeredo Alves Antunes, Professor Lívia Azeredo Alves Antunes, Universidade Federal Fluminense
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDI treatment and OHRQoL
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Trauma Dental; Quality of Life
Keywords: oral heath; quality of life; tooth injuries; children; family
MeSH Terms: conditions — Tooth Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TDI treatment (Experimental): The TDI treatment was performed according to its complexity. Uncomplicated TDI received minimally invasive treatment (simple restorations and clinical and radiographic follow-up). Complicated TDI received invasive treatment (more complex restorations, endodontic treatment, confection of aesthetic devices, restraints).
  The Oral Health Related to Quality of Life assessment will be conducted before treatment (Baseline) and from between 3 to 6 months after the TDI treatment .
  Interventions: Procedure: TDI treatment

INTERVENTIONS:
Procedure: TDI treatment — The TDI treatment was performed according to its complexity. Uncomplicated TDI received minimally invasive treatment (simple restorations and clinical and radiographic follow-up). Complicated TDI received invasive treatment (more complex restorations, endodontic treatment, confection of aesthetic devices, restraints).

SUMMARY:
The aim of this research was to assess the impact of Oral Health-Related Quality of Life (OHRQoL) on children and their families affected by Traumatic Dental Injury (TDI) after insertion into a Dental Trauma Care Program (DTCP). After a sample size calculation, this non-randomized clinical study was composed of a consecutive sample of 2 to 6-year-old children registered in the DTCP from 2012-2019. Parents/Caregivers were interviewed to fill up an OHRQoL questionnaire. The Brazilian version of the Early Childhood Oral Health Impact Scale (B-ECOHIS) was applied (in form of an interview) to evaluate the impact of TDI on OHRQoL before, and after treatment. The scores of the B-ECOHIS were calculated using the additive method, summing the numeric response codes for each item. The Andreassen classification was used to determine the TDI. The patients were treated (minimally intervention/invasive intervention) according to TDI severity (uncomplicated/complicated). The Kolmogorov-Smirnov test was performed to evaluate the normality of the data to determine the use of parametric or non-parametric tests. Mean or median comparisons were made for items in the overall scale and subscale scores to compare B-ECOHIS total scale/subscales/domains before and after insertion in DTCP. The responsiveness was assessed by analyzing the change in the scores on the scales and subscales. The changes were calculated by subtracting the post-treatment scores from the before-treatment scores. Positive change scores indicate an improvement in OHRQoL, while negative scores indicate deterioration. TDI severity and treatment-associated were also evaluated.

DETAILED DESCRIPTION:
It is recognized that measurements OHRQoL are essential strategies of oral health surveys, clinical trials, and studies evaluating the outcomes of preventive and therapeutic program. In the literature it is observed efficacy on OHRQoL outcomes focused on oral health education (OHE) associated to: atraumatic restorative treatment (ART), dental caries, gingivitis.

In the literature it is also seen that the presence of TDI is associated to negative impact on OHRQoL)that affects physical and psychosocial consequences for children and their families. The treatment of TDI is a challenge, that it is related to an improvement on famil and on children from 8 to 14 years and attended in a center of surveillance for TDI.

For a broader understanding of the consequences of outcomes of preventive and therapeutic program for TDI, it is important to expand the assessment of its performance using an OHRQoL measure for other ages of children.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 2 to 6 years who suffered some type of TDI in the deciduous dentition
* healthy patients without disabilities
* children don't used interceptive orthodontic braces or prostheses
* TDI that occurred in the last 3 months before the first questionnaire application
* TDI treatment completed up to 3 months before the second questionnaire application

Exclusion Criteria:

* parents/caregivers that refuse to answer the questionnaire at any point
* parents/caregiversor who do not agree to sign the consent terms

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Impact on oral heath related to quality of life from children and their families affected by traumatic dental injuries evaluated by B-ECOHIS instrument | 6 months
  The B-ECOHIS was applied (in form of interview). This questionnaire is composed of 13 items distributed between a child impact section (CIS) and family impact section (FIS). The first section has four subscales: symptoms, function, psychology and self-image/social interaction. The FIS has two subscales: parental distress and family function. Response categories of ECOHIS were coded on a five-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = often; 4 = very often. All 'don't know' responses were recoded to "never". The score for each domain is calculated through a simple sum of the scores of each item. The total score ranges from 0 to 52. After the TDI treatment a follow-up will be performed. The changes were calculated by subtracting the appointment 2 (follow up) from the appointment 1 (initial exam). Positive change scores indicate an improvement in OHRQoL, while negative scores indicate deterioration.

SECONDARY OUTCOMES:
Impact on oral heath related to quality of life from children and their families affected by traumatic dental injuries according TDI severity and type of TDI treatment evaluated by B-ECOHIS instrument | 6 months
  The B-ECOHIS was applied (in form of interview)and was used to evaluate the impact of the TDI according to its severity (complicated or uncomplicated) and type of treatment (minimally invasive or invasive). This questionnaire is composed of 13 items distributed between a child impact section (CIS) and family impact section (FIS). The first section has four subscales: symptoms, function, psychology and self-image/social interaction. The FIS has two subscales: parental distress and family function. Response categories of ECOHIS were coded on a five-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = often; 4 = very often. All 'don't know' responses were recoded to "never". The score for each domain is calculated through a simple sum of the scores of each item. The total score ranges from 0 to 52, with higher scores denoting greater oral health impact and poorer OHRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Livia A Antunes, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil